CLINICAL TRIAL: NCT05832723
Title: A Real-world Study to Evaluate the Efficacy of 650nm Low-intensity Single-wavelength Red Light in the Prevention and Control of Myopia in Children and Adolescents
Brief Title: A Real-world Study of 650nm Low-intensity Single-wavelength Red Light for Children and Adolescents
Status: Recruiting | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Ying Jie, MD, Prof, Beijing Tongren Hospital
Other Study IDs: TongrenJY2023
Record Dates: First submitted 2023-03-19; First posted 2023-04-27 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 650 nm low-level red-light: Children who are exposed to the 650 nm low-level red-light will be recruited into the cohort, the exposure factor is red-light irradiation. The study does not give interventions, but only recruit children who received or who is receiving the 650 nm low-level red-light intervention for observation.
  Interventions: Device: 650 nm low-level red-light

INTERVENTIONS:
Device: 650 nm low-level red-light — Typically, children who uses the 650 nm low-level red-light will be recruited into this study. The use of any other myopia intervention is not restricted except for low concentrations of atropine. Because atropine will cause pupils dilated, the amount of light entering the eye can not be controlled, and red-light is a laser, to be safe, we need to take certain consideration of the amount of light-entering. Participants receive the 650 nm low-level red-light intervention not because they are enrolled in a study, they would receive the intervention in the same manner and intensity if they were not enrolled in the study.

SUMMARY:
To evaluate the efficacy and safety of 650nm low-level red-light irradiation for myopia control and prevention in children under less restrictive conditions than randomized controlled trials. Participants included children(aged 7 to 18 years, spherical equivalent error of 0.5D or below) who are already myopic at recruitment, and those who are of Emmetropia or low hyperopia.

DETAILED DESCRIPTION:
This multicenter real world study will be conducted in at least 100 hospitals: Beijing Tongren Hospital will be the initiator of the study, other hospitals such as the Capital Institute of Pediatrics will serve as sub-centers. The whole study will last for three years.The investigators will perform data analysis at 6 months follow-up, one-year follow-up, and two-year follow-up. Participants who used 650 nm low-level red-light would be recruited. This kind of intervention will be integrated into a headworn device. This device could be used for treatment of myopia or amblyopia, and is safe for the eyes and has been verified by the Chinese market supervision and administration department.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7 to 18 years
2. The cycloplegic spherical equivalent error (SER) is +0.5D or less in both eyes
3. Astigmatism of 2.5 D or less (≤2.5D)
4. Willing to participate in the study and sign the informed consent form

Exclusion Criteria:

1. Including but not limited to the following eye diseases: strabismus, amblyopia, ocular tumors, glaucoma/macular disease and other fundus diseases (including heredity), keratitis, eye trauma, uveitis
2. Including but not limited to the following systemic diseases: epilepsy, tumor, heart disease, asthma, systemic immune diseases, infectious diseases
3. Mental diseases
4. Similar interventions have been used in the past year
5. Allergic to cycloplegic agents or to red light
6. The 650nm red light intervention was not suitable for the condition evaluated by the researchers
7. are currently using atropine or similar drugs, or have stopped using them for less than 1 month

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 7-18 years, and is willing to use 650 nm low-level red-light to control or prevent myopia.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2026-03-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in axial length | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an optical biometer to measure the axial length
Change in spherical equivalent error | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Children's pupil were dilated using Mydrin-P eye drops, and then the refractive error was measured using an autorefractor. the two measurements (axial length and spherical equivalent error) will be aggregated to arrive at one reported value through the following way: axial enlongation will be defined as progress in myopia, decrease in spherical equivalent error will be defined as progress in myopia too.

SECONDARY OUTCOMES:
Change in Choroid thickness to measure | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an enhanced-depth imaging technique (based on Optical coherence tomography )
Change in steep keratometry | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an optical biometer to measure
Change in flat keratometry | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an optical biometer to measure
Change in length thickness | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an optical biometer to measure
Change in anterior chamber depth | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an optical biometer to measure
Change in central corneal thickness | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Use an optical biometer to measure

OTHER OUTCOMES:
Fundus injury related to 650 nm low-level red-light irridiationexamination | Baseline, six-month follow-up, one-year follow-up, two-year follow-up
  Any potential fundus injury related to 650 nm low-level red-light irridiation would be checked through Fundus photography and coherence tomography examination

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jie, PhD, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Red light, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No